CLINICAL TRIAL: NCT02734160
Title: A Phase 1b Dose-Escalation and Cohort-Expansion Study of the Safety, Tolerability, and Efficacy of a Novel Transforming Growth Factor-β Receptor I Kinase Inhibitor (Galunisertib) Administered in Combination With the Anti-PD-L1 Antibody Durvalumab (MEDI4736) in Recurrent or Refractory Metastatic Pancreatic Cancer
Brief Title: A Study of Galunisertib (LY2157299) and Durvalumab (MEDI4736) in Participants With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15784; H9H-MC-JBEG (Other: Eli Lilly and Company); 2015-005295-26 (EudraCT Number)
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08-01

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: immunotherapy; check point inhibitors; transforming growth factor (TGF)-beta R1 kinase inhibitor
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — LY-2157299; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Galunisertib + Durvalumab (Experimental): (Dose Escalation and Cohort Expansion) Galunisertib administered orally in combination with durvalumab administered intravenously (IV).
  Interventions: Drug: Galunisertib; Drug: Durvalumab

INTERVENTIONS:
Drug: Galunisertib — Administered orally
  Other Names: LY2157299
Drug: Durvalumab — Administered IV
  Other Names: MEDI4736

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of the study drug known as galunisertib administered in combination with the anti-programmed cell death-ligand 1 (PD-L1) antibody durvalumab in participants with refractory metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologic or cytologic confirmation of recurrent metastatic pancreatic adenocarcinoma based on standard diagnostic criteria. Recurrence must be documented by diagnostic biopsy.
* Have measurable disease as defined by Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
* Have had disease progression, been refractory or intolerant to no more than 2 prior systemic regimens for locally advanced or metastatic pancreatic cancer. Participants who have received prior neoadjuvant therapy and who now have metastatic disease must have received 1 of the following for their metastatic disease: FOLFIRINOX, nanoparticle albumin-bound paclitaxel/gemcitabine, TS-1 (tegafur gimeracil oteracil potassium), irinotecan liposome injection/5-fluorouracil (5FU)/Leucovorin or single-agent gemcitabine prior to enrolment in this study.
* Dose Escalation: Able and willing to give valid written consent to undergo a new tumour biopsy (prior to study treatment) or to provide an available archival tumour sample if taken <3 years prior to enrolment if a new tumour biopsy is not feasible with an acceptable clinical risk.
* Cohort Expansion: Able and willing to give valid written consent to undergo a new tumour biopsy (prior to study treatment). Able and willing to undergo a second tumour biopsy on treatment. Where possible, tumour lesions used for new biopsies should not be the same lesions used as RECIST target lesions, unless there are no other lesions suitable for biopsy. Archival samples may be required if there is inadequate tissue in the biopsy specimen.
* Have adequate organ function.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Use approved contraceptive methods.

Exclusion Criteria:

* Have moderate or severe cardiovascular disease:

  * Have the presence of cardiac disease, including a myocardial infarction within 6 months prior to study entry, unstable angina pectoris, New York Heart Association Class III/IV congestive heart failure, or uncontrolled hypertension.
  * Have documented major electrocardiogram (ECG) abnormalities (not responding to medical treatments; for example, atrial fibrillation, bundle branch blocks, or as approved by the sponsors).
  * Have major abnormalities documented by ECHO with Doppler (for example, moderate or severe heart valve function defect including moderate or severe valve stenosis or regurgitation, left ventricular ejection fraction <50%, evaluation based on the institutional lower limit of normal, septal aneurysm or other heart aneurysm, any aneurysm of the major vessels or any condition that results in increased risk of aneurysm (eg, Marfan syndrome, patent foramen ovale [PFO]).
  * Have predisposing conditions that are consistent with development of aneurysms of the ascending aorta or aortic stress (for example, family history of aneurysms, Marfan syndrome, PFO, bicuspid aortic valve, evidence of damage to the large vessels of the heart documented by computerized tomography [CT] scan with contrast or magnetic resonance imaging [MRI]).
* Have evidence of interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity or active, noninfectious pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Galunisertib in Combination with Durvalumab Dose-Limiting Toxicities (DLTs) | Cycle 1 (28 Days)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of Galunisertib | Predose Day 1 Cycle 1 through Predose Day 1 Cycle 7 (28 Day Cycles)
PK: Area Under the Curve (AUC) at Steady State of Galunisertib | Predose Day 1 Cycle 1 through Predose Day 1 Cycle 7 (28 Day Cycles)
PK: Minimum Concentration (Cmin) of Durvalumab | Predose Day 1 Cycle 1 through Predose Day 1 Cycle 7 (28 Day Cycles)
Number of Participants with Anti-Durvalumab Antibodies | Predose Day 1 Cycle 2 through Predose Day 1 Cycle 4 (28 Day Cycles)
Progression-free Survival (PFS) | Baseline to Objective Progressive Disease or Death (Estimated up to 18 Months)
Objective Response Rate (ORR): Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) | Baseline to Objective Progressive Disease (Estimated up to 18 Months)
Duration of Response (DoR) | Date of CR or PR to Date of Objective Progressive Disease or Death Due to Any Cause (Estimated up to 18 Months)
Disease Control Rate (DCR): Percentage of Participants With a Best Overall Response of CR, PR, and Stable Disease (SD) | Baseline to Objective Progressive Disease or Start of New Anti-Cancer Therapy (Estimated up to 18 Months)
Time to Response | Baseline to Date of CR or PR (Estimated up to 4 Months)
Overall Survival (OS) | Baseline to Date of Death from Any Cause (Estimated up to 30 Months)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- United States (4):
  - Honor Health Research Institute, Scottsdale, Arizona
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
- Gustave Roussy, Villejuif, France
- Ospedale Policlinico Giambattista Rossi, Borgo Roma, Verona, Italy
- South Korea (2):
  - Samsung Medical Center, Seoul, Korea
  - Seoul National University Hospital, Seoul
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid

REFERENCES:
- [Derived] Melisi D, Oh DY, Hollebecque A, Calvo E, Varghese A, Borazanci E, Macarulla T, Merz V, Zecchetto C, Zhao Y, Gueorguieva I, Man M, Gandhi L, Estrem ST, Benhadji KA, Lanasa MC, Avsar E, Guba SC, Garcia-Carbonero R. Safety and activity of the TGFbeta receptor I kinase inhibitor galunisertib plus the anti-PD-L1 antibody durvalumab in metastatic pancreatic cancer. J Immunother Cancer. 2021 Mar;9(3):e002068. doi: 10.1136/jitc-2020-002068. PMID 33688022
- See also: Click here for more information about this study: A Study of Galunisertib (LY2157299) and Durvalumab (MEDI4736) in Participants With Metastatic Pancreatic Cancer — http://www.lillytrialguide.com/en-US/studies/pancreatic-cancer/JBEG#?postal=